CLINICAL TRIAL: NCT04527653
Title: Evaluation of the Efficacy and Safety of a Thermal Fractional Skin Rejuvenation System (Tixel) for the Treatment of Facial and/or Scalp Actinic Keratoses
Brief Title: Evaluation of The Efficacy and Safety of Tixel Treatment for the Treatment of Facial and/or Scalp Actinic Keratoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novoxel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 0732
Record Dates: First submitted 2020-08-17; First posted 2020-08-26 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: Single-center, Prospective, Open Label, with Before-After Study Design
Masking Description: The mean of the improvement in actinic keratosis performed by two independent dermatologists using photograph images taken at baseline and at 4, 12-weeks follow-up visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tixel Treatment (Experimental): This is a non-invasive thermo-mechanical treatment to the scalp and/or face using the Tixel technology
  Interventions: Device: Tixel

INTERVENTIONS:
Device: Tixel — Non-invasive thermo-mechanical treatment

SUMMARY:
Evaluation of the Efficacy and Safety of a thermal fractional skin treatment system (Tixel) for the treatment of facial and/or scalp actinic keratoses

DETAILED DESCRIPTION:
Single-center, Prospective, Open Label, with Before-After Study Design. Up to 25 subjects will be enrolled to the study to provide at least 20 evaluable subjects. Subjects will be examined to determine the severity and extent of actinic keratoses.

All subjects will undergo 1-3 treatments (determined by their clinical improvement), 3-4 weeks apart.

Follow-up visits after the last treatment visit: 4 weeks (±7 days), 12 weeks (±7 days), 52 weeks (±14 days) - the last follow up visit is a voluntary one.

The inclusion criteria would be mild to moderate thickness confluent actinic keratoses located to scalp and/or face.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Skin Photo type I-VI
* Mild to moderate thickness confluent actinic keratoses located to scalp and/or face
* Subject is willing and able to comply with protocol requirements and all study visits
* Subject has provided a written informed consent

Exclusion Criteria:

* Any patient who has undergone tanning during the 4 weeks prior to any treatment session and/or any patient who plans to undergo tanning during the 4 weeks following any treatment session (patients who may be exposed to the sun for short periods of time occasionally are not contra-indicated as long as they apply a high SPF sunscreen (>50).
* Current active Herpes Simplex infection.
* Current skin cancer, malignant sites and/or advanced premalignant lesions or moles in the treatment area.
* An impaired immune system condition or use of immunosuppressive medication.
* Collagen disorders, keloid formation and/or abnormal wound healing.
* Any patient who takes or has taken any medications (including via topical application), herbal treatment (oral or topic), food supplements or vitamins, which may cause fragile skin or impaired skin healing during the last 3 months.
* Any patient who has used oral Isotretinoin (Accutane® or Roaccutan®) within 3 months prior to treatment or less.
* Any patient who has a history of bleeding coagulopathies.
* Any patient who has tattoos or permanent makeup in the treated area.
* Any patient who has burned skin, blistered skin, irritated skin, or sensitive skin in any of the areas to be treated.
* Women who are pregnant (as determined by self-reporting), lactating, or less than 3 months post-delivery, possibly pregnant or planning a pregnancy during the study period.
* Currently participating in or recently participated in another clinical trial (within the last 30 days).
* Age below 18 years.
* Subject underwent prior treatments for actinic keratoses including:
* Prior treatment with ablative laser, any laser or photo-dynamic therapy 3 months prior to enrollment.
* Any cryotherapy or electrodessication 6 weeks prior to enrollment.
* Systemic retinoid therapy within 6 months prior to enrollment.
* Topical treatment with 5-Fluorouracil cream and/or imiquimod cream and/or diclofenac gel and/or ingenol mebutate gel 6 months prior to enrollment.
* Face cannot be treated due to dermal disorder other than actinic keratoses, such as infection, surgical treatment etc.
* Subject has a systemic disease manifested by actinic keratoses (e.g. immune suppression).
* Significant systemic illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Blinded Evaluation of Improvement | 6 months
  lesions count as well as an evaluation of the overall improvement in facial appearance based on a quartile scale of improvement graded as 0 (exacerbation) 1 (1-25% improvement), 2 (26-50% improvement), 3 (51-75% improvement) or 4 (76-100% improvement)]
Safety, number of Adverse Events | 6 months
  Any safety related event during the study will be record and analysed

SECONDARY OUTCOMES:
Subject Satisfaction Assessments | 6 months
  Subjects will assess their satisfaction with the procedure on FU visit. The assessment will be based on a 5-point Likert scale detailed in Table 4 where 0 represents "very dissatisfied" and 4 represents "very satisfied".
Downtime Assessment | 4 moths
  Subject will report the period of time following the procedure during which they had expected side effects
Discomfort Assessment | 3 months
  Subject will assess their pain level following each treatment via Pain Visual Analogue Scale (VAS), were 0 is "no pain" and 10 is "intolerable pain".
Expected immediate response | 3 months
  Investigator will assess expected immediate response and will document immediately post treatment using a 4-level scale: (0) None / (1) Mild / (2) Moderate / (3) Severe on each treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Assi Levi, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Ha'Sharon Campus, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided